CLINICAL TRIAL: NCT00051831
Title: A Pilot Study to Measure the Clearance of Replication-Competent HIV-1 in Resting Memory CD4+ Cells in HIV-1-Infected Subjects Who Receive Enfuvirtide Plus Oral Combination Antiretroviral Therapy
Brief Title: Effect of an Enfuvirtide-based Anti-HIV Drug Regimen on Latent HIV Reservoirs in Treatment Naive Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Advancing Clinical Therapeutics Globally for HIV/AIDS and Other Infections (Network)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A5173; 10006 (Registry Identifier: DAIDS ES); ACTG A5173
Record Dates: First submitted 2003-01-16; First posted 2003-01-20 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Treatment Naive; HIV-1; Virus Replication; CD4-Positive T-Lymphocytes; Immunologic Memory; Pentafuside; Anti-HIV Agents; Drug Therapy, Combination; Saquinavir; Ritonavir; Tenofovir Disoproxil Fumarate; RNA, Viral; Viral Load; Fusion Inhibitors; Entry Inhibitors
MeSH Terms: conditions — HIV Infections | interventions — Emtricitabine; Enfuvirtide; Ritonavir; Saquinavir; Tenofovir

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Emtricitabine; Drug: Enfuvirtide; Drug: Ritonavir; Drug: Saquinavir; Drug: Tenofovir disoproxil fumarate

INTERVENTIONS:
Drug: Emtricitabine — Will be administered as one 200-mg capsule orally daily
  Other Names: FTC; Emtriva
Drug: Enfuvirtide — Will be administered as a 90-mg (1.0 mL) subcutaneous injection twice daily
  Other Names: ENF; Fuzeon; T-20
Drug: Ritonavir — Will be administered as one 100-mg capsule orally twice daily
  Other Names: RTV; Norvir
Drug: Saquinavir — Will be administered as five hard gel capsules orally twice daily
  Other Names: Invirase; Saquinavir mesylate
Drug: Tenofovir disoproxil fumarate — Will be administered as one 300-mg tablet orally daily
  Other Names: TDF; Viread

SUMMARY:
HIV replication in resting CD4 cells is so minimal that anti-HIV drugs often fail to destroy the virus in these cells. Enfuvirtide, also known as T-20, is a type of anti-HIV drug called a fusion inhibitor. The purpose of this study is to test the ability of a T-20-enhanced treatment regimen to decrease the number of resting CD4 cells that become infected with HIV.

DETAILED DESCRIPTION:
While current HIV treatment with combination antiretroviral therapy (ART) has reduced morbidity and mortality, it does not eradicate or cure HIV infection. A possible explanation for this failure is the persistence of virus in long-lived reservoirs. Resting memory CD4 cells have been proposed as providing a cellular reservoir. Most patients who initiate ART during chronic HIV-1 infection do not experience a detectable reduction in HIV in the latent reservoir; this may be due to low levels of ongoing viral replication that maintains the resting CD4 cell reservoir. Increasing the potency of therapy by inhibiting new viral targets may result in a decrease in the number of latently infected cells and clearance of the latent reservoir. Addition of the fusion inhibitor T-20 to ART including reverse transcriptase inhibitors and protease inhibitors (PIs) may help achieve this goal. This study will evaluate whether treatment naive, chronically infected HIV patients treated with T-20 plus emtricitabine (FTC), ritonavir (RTV), saquinavir (SQV), and tenofovir disoproxil fumarate (TDF) have a measurable decline in the latently infected CD4 cell reservoir. Patients and their physicians may choose different PIs than RTV and SQV, but they will not be provided by the study.

Patients in this study will receive injections of T-20 twice daily in addition to oral FTC and TDF once daily and oral RTV and SQV twice daily. At Week 24, patients will have their latent cell reservoir sampled. Patients whose HIV viral loads are less than 50 copies/ml at or after Week 24 but prior to Week 48 will continue the treatment regimen through the end of the study; their latent cell reservoirs will be tested at Weeks 48, 72, and 96. Patients whose viral loads are between 50 copies/ml and 200 copies/ml will continue the treatment regimen and latent cell sampling, but their regimens may be intensified as determined by the study team. Patients whose viral loads are 200 copies/ml or greater after Week 24 may continue their study regimens, but will no longer contribute latent cell samples.

This study will last 96 weeks. During the first 4 months of the study, patients will have 7 study visits; after that, study visits will be every 8 weeks until the end of the study. Medical history, clinical assessments, and blood collection will occur at every study visit. Pill and ENF vial counts will be assessed, and patients will be asked to complete a medication adherence questionnaire at selected study visits.

ELIGIBILITY:
Inclusion Criteria

* HIV-1 infected
* Viral load of 1,000 copies/ml or greater within 60 days prior to study entry
* CD4 count of 100 cells/mm3 or greater within 60 days prior to study entry
* Willing to use acceptable methods of contraception

Exclusion Criteria

* Previous treatment with any nucleoside analogue, nonnucleoside reverse transcriptase inhibitor, or fusion inhibitor for longer than 7 days
* Any previous treatment with T-20, lamivudine, or FTC
* HIV-related vaccine within 6 months prior to study entry
* Evidence of HIV seroconversion within 6 months prior to study entry
* Acute AIDS-defining opportunistic infection (OI). Patients who are not clinically stable or who have not been on therapy for the OI for at least 30 days prior to study entry are excluded. Patients who have no evidence of active disease and have been receiving maintenance therapy for AIDS-related OI for at least 30 days are not excluded.
* Systemic chemotherapy within 30 days of study entry or anticipated need for systemic chemotherapy before the end of the study
* Treatment with immune modulators such as systemic steroids, IL-2, alpha interferon, G-CSF, erythropoietin, or any investigational agent within 30 days of study entry
* Allergy to study drugs or their formulations
* Serious illness, substance abuse, or other medical condition that would compromise the patient's ability to participate in the study
* Certain primary resistance HIV mutations
* Pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2003-10; Primary Completion 2007-12 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Frequency of latently infected CD4+ T cells from peripheral blood with replication-competent HIV-1 (in infectious units per million cells) | Throughout study

SECONDARY OUTCOMES:
Any Grade 3 or 4 adverse experience, including Grade 3 or 4 laboratory value, sign or symptom, and all deaths. | Throughout study
Targeted events and toxicities will also be considered and these include injection site reactions (any grade), bacterial pneumonia, cellulitis | Throughout study
- Level of HIV-1 RNA in plasma as measured by the Roche Ultrasensitive assay | Throughout study
- Level of HIV-1 DNA in PBMC | Throughout study
- Frequency of 2-LTR in PBMC | Throughout study
-Sequence of HIV env and HIV pol genes | Throughout study
-CD8/CD38 antibody binding capacity (ABC) | Throughout study
- Level of HIV-1 RNA in cerebrospinal fluid | Throughout study
- Level of HIV-1 RNA in genital fluid | Throughout study
- Level of HIV-1 RNA in plasma as measured by an ultra-ultrasensitive assay | Throughout study
- Measures of cell surface density of chemokine (CCR5, CXCR5) receptors | Throughout study
- Responses to subject preferences and injection administration concerns questionnaires | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Joseph J. Eron, Jr., MD, Study Chair — University of North Carolina, Chapel Hill
Locations (7):
- United States (6):
  - University of Colorado Hospital CRS, Aurora, Colorado
  - Massachusetts General Hospital ACTG CRS, Boston, Massachusetts
  - Washington U CRS, St Louis, Missouri
  - NY Univ. HIV/AIDS CRS, New York, New York
  - Unc Aids Crs, Chapel Hill, North Carolina
  - The Ohio State Univ. AIDS CRS, Columbus, Ohio
- Puerto Rico-AIDS CRS, San Juan, Puerto Rico

REFERENCES:
- [Background] Blankson JN, Persaud D, Siliciano RF. The challenge of viral reservoirs in HIV-1 infection. Annu Rev Med. 2002;53:557-93. doi: 10.1146/annurev.med.53.082901.104024. PMID 11818490
- [Background] Perelson AS, Essunger P, Cao Y, Vesanen M, Hurley A, Saksela K, Markowitz M, Ho DD. Decay characteristics of HIV-1-infected compartments during combination therapy. Nature. 1997 May 8;387(6629):188-91. doi: 10.1038/387188a0. PMID 9144290
- [Background] Pierson T, McArthur J, Siliciano RF. Reservoirs for HIV-1: mechanisms for viral persistence in the presence of antiviral immune responses and antiretroviral therapy. Annu Rev Immunol. 2000;18:665-708. doi: 10.1146/annurev.immunol.18.1.665. PMID 10837072
- [Background] Kilby JM, Hopkins S, Venetta TM, DiMassimo B, Cloud GA, Lee JY, Alldredge L, Hunter E, Lambert D, Bolognesi D, Matthews T, Johnson MR, Nowak MA, Shaw GM, Saag MS. Potent suppression of HIV-1 replication in humans by T-20, a peptide inhibitor of gp41-mediated virus entry. Nat Med. 1998 Nov;4(11):1302-7. doi: 10.1038/3293. PMID 9809555
- [Derived] Gandhi RT, Bosch RJ, Aga E, Albrecht M, Demeter LM, Dykes C, Bastow B, Para M, Lai J, Siliciano RF, Siliciano JD, Eron JJ; AIDS Clinical Trials Group A5173 Team. No evidence for decay of the latent reservoir in HIV-1-infected patients receiving intensive enfuvirtide-containing antiretroviral therapy. J Infect Dis. 2010 Jan 15;201(2):293-6. doi: 10.1086/649569. PMID 20001856